CLINICAL TRIAL: NCT03259646
Title: The IPV Provider Network: Engaging the Health Care Provider Response to Interpersonal Violence Against Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Office of Research on Women's Health (ORWH) (NIH); University of Pittsburgh (Other); Futures Without Violence (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00090497; 6 ASTWH150032-01 (Other Grant/Funding Number: Office of Women's Health)
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Violence, Domestic; Violence, Sexual
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Intervention Model Description: cluster randomized trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Universal Education (Experimental): Train providers to integrate screening, universal education, trauma informed counseling, and mobile health (mHealth) technology through the myPlan app safety decision aid in collaboration with local IPV programs as well as the integration of documentation and quality improvement templates and measures into clinical settings.
  Interventions: Behavioral: Universal Education
- Standard Practice (No Intervention): Standard clinical practice

INTERVENTIONS:
Behavioral: Universal Education — Clinic provider/staff training on implementing universal education into clinical practice to: 1.) provide all women information about IPV/SA, harm reduction, and available safety resources; 2) provide trauma-informed counseling to women who disclose IPV/SA; includes access to the myPlan safety decision aid to develop a tailored safety action plan; 3) provide warm referrals in partnership with local domestic violence and sexual assault (DV/SA) advocacy agencies; 4) integrate documentation and quality improvement templates and measures into clinical settings.
  Arms: Universal Education

SUMMARY:
Violence against women is a major public health threat that carries significant consequences for women's health. Moreover, women experiencing intimate partner violence (IPV) and sexual assault (SA) are more likely than non-abused women to seek certain forms of health services, such as for sexually transmitted infections, chronic pain and illnesses, depression and/or pregnancy-related concerns. As a result, the health sector is an ideal setting to identify and support survivors. The U.S. Institute of Medicine has identified the health care system, including the public health infrastructure, as key for identification of and support for survivors of violence, as well as for violence prevention. While some evidence-based models exist, no current national consensus has been reached on scalable best practices in screening and brief counseling for IPV/SA.

This multi-level intervention includes integrating into the clinic setting IPV/SA screening, universal education, trauma informed counseling, warm referrals (e.g. provider/staff contact advocacy program with survivor) to local IPV/SA advocacy agencies, and access to the evidence-based myPlan safety decision aid app. The evaluation, using a cluster randomized trial design, will measure longitudinal outcomes (over 6 months) of patient self-efficacy, health and safety outcomes, as well as participant and provider perceptions of the intervention and clinic level changes in primary and reproductive health clinics in four states (Arizona, Massachusetts, Pennsylvania and West Virginia) to achieve the following aims:

Aim 1. Evaluate the effectiveness of an evidence-based screening, universal education and trauma-informed counseling with tailored safety action plan and referrals to partner IPV/SA programs compared to standard practice, on survivor health and safety outcomes over a cumulative period of six months.

Aim 2. Examine longitudinal changes in clinic-level screening, universal education, trauma informed counseling, safety action plans and referrals to on-site and/or partner IPV/SA programs and improved standards for documentation through the electronic health record (EHR) and continuous quality measurement and reporting.

ELIGIBILITY:
Inclusion Criteria:

* Seeking healthcare at one of 14 partner clinics
* Ability to complete a survey on a device (computer/tablet/smartphone in English or Spanish)
* Access to safe device (as defined above) if doing surveys online
* Has a safe email address or safe phone number
* Is not acutely ill

Exclusion Criteria:

* Male
* Not seeking healthcare at one of 9 partner clinics
* Younger than 18 years of age
* Older than 59 years of age
* Cannot read/speak English or Spanish
* No access to safe device if doing surveys online
* Does not have a safe email address or safe phone number
* Acutely ill

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cis-gender or trans-gender women.
Enrollment: 6272 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Change in use of safety behaviors | 6 months
  Measured by percent of safety behaviors the woman has tried and found helpful on the Safety Behaviors Checklist. The checklist was adapted from Sullivan and colleagues and Parker and colleagues. Includes use of community resources and safety steps (e.g. asked for help, hidden emergency money) and use of formal services (e.g., women's shelter, protection order, mental health services).
Change in Self-Efficacy to Use Harm Reduction Strategies | 6 months
  Measure adapted from Tancredi et al and Hibbard et al, assesses confidence to seek help for abuse, if needed, from a health care provider.
Provider Behavior | Baseline
  Clinic level measure. Provider Behavior at Visit Survey items administered after the provider visit to assess the provider's adherence to universal education intervention, i.e. discussing healthy and unhealthy relationships during the visit, and referring to resources.

SECONDARY OUTCOMES:
Change in decisional conflict | 6 months
  We have adapted questions from validated subscales of the Decisional Conflict Scale as a measure of decision process. Measures whether the intervention helps a woman to understand the advantages and disadvantages of safety planning options and to know her values related to them. The Decisional Conflict Scale discriminates between people who make decisions and those who delay making decisions.
Change in Readiness to Take Action | 6 months
  0-10 scale of readiness to make changes to relationship for safety

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Glass, PhD, MPH, RN, Principal Investigator — Johns Hopkins University
Locations (9):
- United States (9):
  - North County HealthCare, Kingman, Arizona
  - North Country HealthCare, Lake Havasu City, Arizona
  - North Country HealthCare, Williams, Arizona
  - Partners Health Care Brigham and Women's Hospital, Boston, Massachusetts
  - Magee-Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Women's Health Center, Charleston, West Virginia
  - Valley Health, Mill Creek, West Virginia
  - Greenbrier Co. Health Dept, Ronceverte, West Virginia
  - FamilyCare Health Center, Scott Depot, West Virginia

IPD SHARING:
Plan to Share IPD: No